CLINICAL TRIAL: NCT00238823
Title: A Review and Comparison of Cryoablation and Radiofrequency Ablation in Children
Brief Title: Cryoablation Versus Radiofrequency Ablation
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-108
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2007-05-23 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: cryoablation; radiofrequency ablation; pediatrics; cardiology
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The purpose of this retrospective study is to describe why and when we used cryo and why we crossed over when we used both RFA and cryo. It is also to determine if there is some predictor that would make us say one patient would be better served with one technique than another and to describe our overall acute success rate and then our 6-month recurrence rate with cryo ablation and compare it to our known success rate with RFA.

DETAILED DESCRIPTION:
Cryotherapy (Cryo) is a new ablation energy source used instead of the radiofrequency (RFA) method for ablation of septal pathways. In the past year, we have used cryo approximately 50 times, however 50% of the cryo procedures crossed over from RFA to cryo or cryo to RFA. It appears to me that cryo use should be as an adjunct therapy to RFA instead of replacement of RFA.

I would like to describe why and when we used cryo and why we crossed over when we used both RFA and cryo. I would like to determine if there is some predictor that would make us say one patient would be better served with one technique than another. I would also describe our overall acute success rate and then our 6-month recurrence rate with cryo ablation and compare it to our known success rate with RFA. All of this can be done with a chart review.

This will be done through a retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* charts between January 1 and 2004 to December 31, 2004
* pediatric population
* those who were ablated

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2004-01; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Strieper, DO, Principal Investigator — Sibley Heart Center
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States